CLINICAL TRIAL: NCT05387174
Title: Nursing Intervention in Two Risk Factors of the Metabolic Syndrome, Abdominal Obesity and Arterial Hypertension, and Quality of Life in the Climacteric Period
Brief Title: Nursing Intervention in Two Risk Factors of the Metabolic Syndrome and Quality of Life in the Climacteric Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Concepcion (Other)
Collaborators: Universidad Central del Ecuador (Other)
Responsible Party: Principal Investigator, Alide Salazar Molina, Research Director, Universidad de Concepcion
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEBB 649-2020
Record Dates: First submitted 2022-05-09; First posted 2022-05-24 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Obesity, Abdominal; Hypertension; Quality of Life; Menopause
Keywords: Metabolic syndrome, Menopause, Quality of life
MeSH Terms: conditions — Obesity, Abdominal; Hypertension; Metabolic Syndrome | interventions — Methods; Quality of Life

STUDY DESIGN:
Intervention Model Description: Parallel: participants are assigned to one of two or more groups in parallel for the duration of the study.
Who Masked: Care Provider
Masking Description: As blinding is an unavoidable condition in this type of study, the surveyors in the data collection will not have knowledge about the experimental group and comparison group, so they will be given as group A and B, both at the beginning and at the end of the study in the pre- and post-tests, with the aim of preventing certain biases in some of the stages of the trial and thus protect the sequence after the allocation for convenience.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group nursing intervention with technological support (Experimental): Experimental group composed of 40 with the same characteristics as above and attending the San Antonio de Pichincha Health Center, this group will additionally receive a nursing intervention of 3 months, to reduce the risk factors of MS and improve the quality of life related to health. The nursing intervention with web application support will consist of three elements: Individual face-to-face individual Nursing Counseling, Group Education and Physical Activity sessions through virtual platform.
  Interventions: Behavioral: : Nursing intervention in two risk factors of the Metabolic Syndrome, abdominal obesity and arterial hypertension and quality of life in the climacteric period.
- Group compared regular care at the MSP Health Center (No Intervention): Comparison group composed of 40 women in the climacteric stage between 40 and 59 years old who have two risk factors of MS (abdominal obesity and arterial hypertension), who go to the Health Center of the People's Committee, to the group of the Hypertensive Program that receive the usual attention of the Institution on group talks, health fairs based on general topics of the disease.

INTERVENTIONS:
Behavioral: : Nursing intervention in two risk factors of the Metabolic Syndrome, abdominal obesity and arterial hypertension and quality of life in the climacteric period. — Nursing intervention with technological support (Metamorphosis) in two risk factors of Metabolic Syndrome, abdominal obesity and hypertension and quality of life in the climacteric period, developed in 3 months, in the experimental group that includes individual nursing counseling, group education virtually and physical activity sessions for 12 weeks virtually.
  Arms: Experimental group nursing intervention with technological support

SUMMARY:
The estrogenic deficit characteristic of the climacteric stage is accompanied by a high incidence of health problems, such as the presence of Metabolic Syndrome risk factors that contribute to the increase of cardiovascular diseases.

Objective: To determine the effect of a nursing intervention based on self-care aimed at improving the control of two metabolic syndrome risk factors (abdominal obesity and arterial hypertension) and health-related quality of life in climacteric women.

Material and methods: Quasi-experimental study, non-equivalent control group design with women between 40 and 59 years old who present two risk factors of the Metabolic Syndrome (abdominal obesity and arterial hypertension) from two type C Health Centers of District 17D03 of Quito, Ecuador. Among one of the conceptual hypotheses, the researchers have Conceptual hypothesis 1: Climacteric women of the experimental group after the intervention of Nursing based on self-care improve two risk factors of MS with respect to those of the comparison group. A sample of 40 women was selected for experimental group and 40 for comparison group. Instruments and measurements: Abdominal Circumference, Blood Pressure, Menopause Rating Scale, International Physical Activity Questionnaire (IPAQ). Women in both groups received the usual care and those in the experimental group received a Nursing Intervention with technological support that included individual face-to-face nursing counseling, group education and physical activity sessions through a virtual platform for 12 weeks. Ethical requirements were considered.

Expected results: It is expected that after the Nursing Intervention based on self-care the women of the experimental group will decrease the parameters of abdominal circumference, blood pressure and improve health-related quality of life.

DETAILED DESCRIPTION:
1. INTRODUCTION 1.1 Presentation and rationale of the problem During the last decade, health needs have been changing, with a significant increase in the life expectancy of the population in general and with it the increase of non- communicable diseases, which threaten the health and development of people, especially in developing countries, being predicted for the year 2050.

The World Health Organization (WHO) considers noncommunicable diseases (NCDs) to be the leading cause of morbidity and mortality worldwide, killing 41 million people each year, which is equivalent to 71% of deaths worldwide. Specifically, among individuals aged 30-69 years, 15 million die each year from this type of disease and more than 85% of these premature deaths occur in low- and middle-income countries. According to WHO projections, annual deaths from noncommunicable diseases will increase to 55 million by the year 2030, which at an economic level will bring consequently a high cost to the countries of the world, constituting one of the greatest challenges facing health systems.

Because of the context presented and the projected data, the 2030 Agenda for Sustainable Development recognizes NCDs as a major obstacle to development, WHO has developed the Global Action Plan for the Prevention and Control of Noncommunicable Diseases 2013-2020 to address them. This is expected to reduce premature deaths by 33% by 2030 through prevention and treatment of these conditions (target 3.4 of the Sustainable Development Goals).

Regarding cardiovascular diseases, it is mentioned that the risk factors that are closely related to them are: causal (hypercholesterolemia, hypertension, diabetes mellitus, smoking and age), predisposing (obesity, sedentary lifestyle, family history, sex and psychosocial factors) and conditional (hypertriglyceridemia, high LDL-oxidized, high prothrombotic factor and microalbuminuria), increasing their suffering.

About predisposing factors, it is necessary to consider that the female population is the most affected by cardiovascular diseases because they have a significantly higher risk of mortality, due to their biological difference as well as the complex interactions of cultural and socioeconomic conditions. In this regard, the researchers must consider that female sex, gender, ethnicity, hormonal changes, onset of menarche, pregnancy, premature birth, presence of pathologies such as gestational hypertension, polycystic ovary and menopause, combined with the epidemiological and demographic transition, which have changed habits and lifestyles, further condition the presence of cardiovascular diseases. In addition, the life expectancy of women worldwide has risen considerably and they spend a third or more of their lives after the climacteric period with some risk factor.

The climacteric stage is a physiologically normal period that should be observed due to the permanent cessation of menstruation, after the disappearance of ovarian activity produced by estrogenic decline, which is found between 45 and 55 years of age, marking the end of reproductive life, experiencing physical and emotional changes, because of a series of endocrinological, biological and clinical processes. The hormonal deficit, typical of this stage, is accompanied by a high incidence of problems in women's health (80% hot flashes, night sweats, sleep disorders, fatigue, and depression), as well as the presence of metabolic risk factors that contribute to the increase of cardiovascular diseases, such as acute myocardial infarction.

In this context, the so-called Metabolic Syndrome or Syndrome X arises, characterized by the presence of abdominal obesity, arterial hypertension (AHT), insulin resistance, glucose metabolism disorders and atherogenic dyslipidemia related to metabolic, vascular, inflammatory, ﬁbrinolytic and coagulation abnormalities.

Studies conducted in several countries worldwide indicate that the prevalence of Metabolic Syndrome is found in 60% of the female population and increases in menopause. Thus, studies have shown a high prevalence of Metabolic Syndrome in pre- and postmenopausal women, according to NCEP/ATPIII criteria, with prevalence's ranging from 26.1 to 50.5%, with Ecuador and South Korea standing out in this last group.

That is why the prevalence of Metabolic Syndrome in the climacteric stage constitutes an entity of high epidemiological impact due to the metabolic changes that modify body composition, verifying an increase in weight, insulin resistance and visceral fat, and changes in lipid metabolism and estrogen deficiency that cause deterioration of endothelial function. In addition to the above, hypertension is another factor present among climacteric women with metabolic syndrome. The increase in blood pressure in patients with MS is mainly due to insulin resistance, which causes three actions in the body: increased bioavailability of endothelial nitric oxide; increased activation of the Renin-Angiotensin-Aldosterone System (RAAS) and the endothelin system; changes in the hormonal milieu and a decrease in the autonomic nervous system. In summary, estrogen deficiency can induce sympathetic hyperactivity and endothelial dysfunction by direct effect on the vessels as well as by age-related deleterious effect on the vascular endothelium.

Clinical and epidemiological studies indicate that middle-aged women have at least one independent risk factor for chronic diseases. With this risk approach, it becomes evident how significant preventive work is, aimed at conrolling, reducing and eliminating the risk factors of the Metabolic Syndrome that can complicate the overall health of women at this stage.

Thus, the approach to abdominal obesity and arterial hypertension is particularly relevant in women in the climacteric stage, since women experience during the climacteric period an increase in weight gain and an increase in abdominal adiposity, being this accumulation of visceral fat the major determinant of MS, which is evidenced in 70% of the female population, primarily due to hypoestrogenemia related to metabolic changes, whose distribution is android type, and due to the decrease in muscle mass secondary to the decrease in physical activity. To this is added the approach to arterial hypertension because its prevalence and incidence exceeds the other risk factors of MS by 55%. As arterial pressure is a modifiable risk factor, interventions have been made to control it to levels below 140 mmHg for the systolic and 90 mmHg for the diastolic, reducing cardiovascular risk by 2 to 3% for each mmHg that the diastolic blood pressure (BP) is reduced (TAD).

In addition, the association between the two components of MS (abdominal obesity and hypertension) and the severity of climacteric symptoms have caused negative consequences for women's health, specifically in the domains of physical and psychological health, leading to a deterioration of HRQOL. It is therefore important to consider in all research, the perception of women about their health status, making them active participants in this process, their assessment and contribution is essential to take preventive and therapeutic measures, adapted to the cultural environment in which they are, in order to provide health services, prevent disability and premature death, increasing the years of healthy life and quality of life during the third of their life. It should be noted that there are few intervention studies that integrate the association between the components of MS and quality of life in climacteric women, demonstrating the need to address these variables.

It is therefore essential to carry out comprehensive interventions, undertaking strategies aimed at the promotion and prevention of pathologies prevalent in the climacteric period, such as the Metabolic Syndrome, to reduce cardiovascular risk. It is here that primary health care plays a transcendent role in the control of risk factors, in this context the prevention activities imply behavioral modifications in which educational intervention, health advice and the use of technologies have been effective resulting in the improvement of the quality of life.

In this scenario, the nursing professional plays a crucial role since studies show the nurse's responsibility in the implementation of strategies to contribute to the control of modifiable risk factors of MS, actively involving women in the participation of their own health status. Among some interventions carried out by nurses, there are motivational and technological programs that included physical activity, adequate nutrition, and individualized counseling in women with MS older than 40 years and postmenopausal, reporting positive results in the increase of health- related quality of life in the woman's life and in the control of MS risk factors. However, the inclusion of health-related quality of life and the use of nursing models and theories to guide interventions has been scarcely visible in this type of studies.

Therefore, the following study question leads to the formulation of the problem: What is the effect of a nursing intervention based on self-care to reduce two components of MS (abdominal obesity, hypertension) and improve health-related quality of life in women in climacteric stage attending primary health care centers in the city of Quito- Ecuador? 1.3 HYPOTHESIS

Conceptual Hypothesis 1:

Climacteric women in the experimental group after the self-care nursing intervention improve two MS risk factors over those in the comparison group.

Working hypothesis:

* Climacteric women in the experimental group have lower abdominal circumference after the self-care-based nursing intervention than those in the comparison group.
* Climacteric women in the experimental group have lower systolic blood pressure after the self-care-based nursing intervention than those in the comparison group.
* Climacteric women in the experimental group have lower diastolic blood pressure after the self-care-based nursing intervention than those in the comparison group.

Conceptual Hypothesis 2: Climacteric women in the experimental group after the self- care-based nursing intervention improve health-related quality of life relative to those in the comparison group.

Working hypothesis:

* Climacteric women in the experimental group show lower somatic dimension scores after the self-care-based nursing intervention than those in the comparison group.
* Climacteric women in the experimental group show lower scores in the psychological dimension after the self-care-based nursing intervention than those in the comparison group.
* Climacteric women in the experimental group show lower scores in the urogenital dimension after the self-care-based nursing intervention compared to those in the comparison group.

Conceptual Hypothesis 3: Climacteric women in the experimental group after the self- care-based nursing intervention improve self-care agency by increasing physical activity relative to those in the comparison group.

Working hypothesis:

• Climacteric women in the experimental group improve their level of physical activity after the self-care-based nursing intervention compared to those in the comparison group.

1.4 GENERAL OBJECTIVE To determine the effect of a Nursing Intervention based on self-care aimed at improving the control of two Metabolic Syndrome risk factors (abdominal obesity and arterial hypertension) and health-related quality of life in climacteric women.

Specific Objectives

Regarding women in climacteric stage with two risk factors of Metabolic Syndrome of the experimental group and comparison:

1. To characterize according to basic conditioning factors, the bio-sociodemographic profile, and the level of physical activity.
2. To assess the need for therapeutic self-care using the two MS risk factors (abdominal obesity and arterial hypertension) and health-related quality of life in a pre- and post-test measurement.
3. To evaluate the effect of the self-care-based nursing intervention in the experimental group versus the traditional approach in the comparison group:

   * Risk factors for MS (abdominal obesity and arterial hypertension).
   * Health Related Quality of Life
   * Physical Activity Level 2 SUBJECTS AND METHODS. 2.1 Study design A quasi-experimental, non-equivalent control group design study will be conducted . This type of design is used when the researchers are trying to demonstrate the efficacy of an intervention, but the random assignment of participants is unfeasible, in the context or logistical conditions of recruitment, as in the case of this study.

Within the requirements of the experimental design are considered:

* The independent variable (nursing intervention) will be applied to the experimental group and the variation in the dependent variables (abdominal circumference, blood pressure and health-related quality of life (primary outcome) and physical activity (secondary outcome) will be studied.
* The effect of the independent variable (nursing intervention) on the dependent variables will be measured.
* For control and internal validity, the two groups (experimental and comparison) that are similar before the intervention should be compared and then the effect of the intervention on the dependent variables will be determined.

Making known:

G: Group of people (G1 group 1, G2 group 2). X: Experimental condition (presence of some level or modality of the independent variable), in this research it will be the nursing intervention.

OR: A measurement of the subjects in a group (application of instruments, measurements). If it appears before the experimental condition, it is a pre-test (pre-intervention). If it appears after the experimental condition, it is a post-test (post- intervention).

2.2 Origin The study will be conducted in District 17D03 of the Ministry of Public Health of Ecuador. This district has two Type C Health Centers: San Antonio de Pichincha Health Center and Comite del Pueblo Health Center. These facilities are part of the National Health System and are in the urban sector, north of the city of Quito. They provide services to a population of 25,000 to 50,000 inhabitants and provide coverage to approximately 13,000 women between the ages of 40 and 59. They offer outpatient services: General Medicine, Gynecology, Pediatrics, Obstetrics, Dentistry, Psychology, Laboratory, Ultrasound, Pharmacy, Nursing, Vaccinations, Statistics and Emergency, Primary Care Programs (Immunizations, Prevention and Control of TB, Hypertensive and Diabetic Program, among others) from 8 am - 15 pm.

The purpose of carrying out the study in these Centers is by the characteristics and similar population number and because within the functions of the centers of Health type C at level of Country is the promotion of the health, prevention of diseases and recovery of the health by cycles of life, through the services of general medicine, gynecology, infirmary, maternity of short stay and emergency. It is worth mentioning that the hypertensive programmers of the health centers meet three times a month and carry out activities aimed at health promotion and disease prevention.

1. st Phase: Intervention Design Construction of the mobile app and content of the intervention It will be designed and developed through the exploration of content necessary for the intervention of the mobile app during the months of April to July 2021, which will serve as support for the nursing counseling modality, included in the intervention. Having a virtual application will allow combining the technological with personalized interventions, whose design approach will focus on the user, ensuring the needs of the participants and their context, making them participants in the process and development of the product.

   For the construction of this mobile app has been considered, in the first term, a search in the scientific literature based on the topics addressed, incorporating elements of the Self-Care Deficit Theory of Orem. Subsequently, to collect information from users in the climacteric stage, an exploration stage will be carried out where women from the Cotocollao Health Center, with similar characteristics to those of the experimental and comparison group, will be invited to participate in individual interviews, prior Informed Consent, to identify their needs. The inclusion criteria to participate in the interviews will be the same as those required for the intervention. A guideline for the interviews will be developed that integrates aspects related to expectations and suggestions on how to approach health care and the use of technology based on questions asked by the thesis candidate.

   Finally, health care providers (nurses, doctors, nutritionist, physical culture teacher) with a long experience in working with women in climacteric stage and women with presence of risk factors of Metabolic Syndrome will be consulted. The professionals will be invited to participate as consultants regarding the content and time of applicability. Among the professionals, the participation of Dr. Peter Chedraui, an expert in topics related to women in the climacteric stage, has been considered. In addition, support will be provided by eHealth experts and information technology (IT) developers, as well as designers and content specialists who will collaborate with the project team with extensive experience in the development of self-management technology tools.

   Once the necessary content adjustments and input from the participants that will be identified in the exploration phase have been obtained, the first version of the low- fidelity software prototype will be developed, which will consist of the paper prototype that will provide a home page, menu page and screens that will present the design of the first intervention module and content.

   In the first meeting with the eHealth experts, they will test and give feedback on the prototype to ensure the logical creation to meet the requirements of the participants, then the researcher will meet with health experts to socialize the contents of the module and give feedback on its development.

   Subsequently, the high-fidelity prototype will be developed which will have the actual software home page, menu page and modules for the intervention, to ensure usability a second meeting will be held with users, health care providers, subject matter experts and eHealth experts to test it and the feedback data will be used to evaluate, refine, adjust, update the prototype, and verify its usability.

   The security, privacy and confidentiality of eHealth data will depend on the operating software, the device, the network and the servers, it is here, that apart from the technology the researchers will address security issues related to the behavior of the user based on her context and the national policy where the Ministerial Agreement 5216 art. 8, 10, 11, 18 of the Ministry of Public Health of Ecuador points out the security and confidentiality of physical and digital data from collection to disposal.

   The data obtained during the execution of the intervention will be eliminated in a period of five years, counting from the moment of the collection of the information, as indicated in Art. 18 of the Organic Law of Transparency and Access to Public Information, to guarantee that there is no risk of exposure. The storage of the data will be carried out in the servers of the Information Technology Department of the UdeC where the files and the database will be stored in the user: metamorphosis; server: www2.udec.cl; service: ftp; with the domain: metamorfosis.udec.cl, for which the respective authorizations are available.

   Design of the implementation plan This plan constitutes the central part of the intervention, as it allows for the development of an implementation plan. To do this, it will be necessary to identify the facilitating factors and barriers to the adoption and implementation of the intervention, which will allow its evaluation for future implementation.

   The technological support will be used by the participants of the experimental group from the beginning of the nursing intervention. The researcher in the first session of individual counseling, will be responsible for downloading and entering the username and password to each participant to access the application, if the user agrees to work with her phone as a means of support, teaching her how to use it.

   Users will use the app to complement face-to-face individual counseling (3 sessions), virtual group education (2 sessions) and virtual physical activity (36 sessions) by providing remote nursing care from primary care to the home, not to mention reducing the cost of traveling to health centers.

   Designing an evaluation plan the researchers will evaluate the achievement of the implementation of the intervention with technological support based on the self-care of women in the climacteric stage who present two risk factors of MS to improve the quality of life. The objective will be to have a cell app that will be downloaded on the cell phones of the participants during the 3 months of the intervention being useful, attractive, motivating, that fits in the broader context of the daily life of women in the climacteric stage with MS risk factors. The implementation of the technology will aim to reduce costs and intensify the support provided to multiple clients to assist in decision making at the primary care level by providing free access to content developed and refined together with the clients, which will expand equitable access to new resources at the community level and may provide the opportunity to make health care more effective, better coordinated, and closer to home.

   According to what has been previously described, a first (virtual) meeting will be held with the physical culture teacher to socialize the physical activity plan and the instrument to be used during the evaluation and subsequent diagnosis of the physical condition of the participants during the month of July. A week after the initial meeting will be requested collaboration of students of physical culture of the 8th semester, these students will not have knowledge of the group to which the participants belong.

   The second face-to-face meeting will be held with the nursing interns to whom the researcher will train in the application of the instruments to be used in the pre- and post-test, as well as in the measurement of anthropometric parameters and vital signs (blood pressure, heart rate, weight, height, BMI, abdominal circumference) in the month of August. These students will not know which group each participant belongs to.

   The operational, economic and technical feasibility of the project will be carried out through the funding of the researcher and the ethical aspects involved, will be safeguarded from the beginning of the study considering the criteria of Ezekiel Emanuel through the confidentiality of data and informed consent providing autonomy to the participants of the experimental and comparison group to decide for themselves whether or not to participate in the research and withdraw when they deem appropriate, indicating the benefits and risks in an equitable manner among potential participants without seeking to produce harm, since the protection of the person is more important than the search for knowledge.
2. nd Phase: Execution of the intervention In first instance the participants of the group comparison that go to the Center of Health of the Committee of the People and that are registered in the Program of Hypertensive will receive habitual attention of the Institution on group chats, fairs of health based on general topics of the disease and group sessions 2 times per week. In the collection of the data for the investigation the group will receive a copy of the anthropometric measures and indicators of health pre, and post intervention and they will continue with their habitual activities.

On the other hand, the participants of the experimental group will receive counseling through: Educational counseling with technological support (3 individual sessions), educational sessions (2 group sessions virtually) and physical activity sessions 3 times a week virtually and an individual walking session. The topics of annual clinical controls, Metabolic Syndrome risk factors, health-related quality of life, healthy eating, and adequate level of physical activity in the climacteric stage will be included, which will be focused on self-care to improve the usual lifestyles. These sessions will be taught by the nurse/researcher.

ELIGIBILITY:
Inclusion Criteria:

* Be between 40 and 59 years of age.
* Abdominal circumference equal to or greater than 80 cm.
* Blood pressure equal to or greater than 130/85mmHg or on antihypertensive treatment
* Being able to ambulate without assistance.
* Population residing in the sector in which you are registered.
* Access to mobile or fixed internet service.

Exclusion Criteria:

* Women on hormone replacement therapy.
* Women with hysterectomy and/or oophorectomy
* Pregnant women.
* Women with cardiovascular disease such as dyslipidemia, type II diabetes; cancer; hypothyroidism; respiratory disease; neuromuscular or terminal illness.
* People who cannot read or write.

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2021-09-11 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Change in abdominal obesity | Until the end of the study (3 months duration)
  Anthropometric measurements (abdominal circumference)
Reduce systolic and diastolic blood pressure | Until the end of the study (3 months duration)
  Vital sign (systolic and diastolic blood pressure)
Improve health-related quality of life | Until the end of the study (3 months duration)
  Instrument Menopause Rating Scale: (Minimum total value "0 points" and maximum "44 points", if the score is higher the result is negative)

SECONDARY OUTCOMES:
Increase the level of physical activity | Until the end of the study (3 months duration)
  International Physical Activity Questionnaire:(Inactive: less than 10 minutes in a row in the last 7 days, Low Activity: between 10 and 149 minutes in the last 7 days and Medium or High Activity: 150 or more minutes in the last 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra C Riofrío Terrazas, Dra (c), Principal Investigator — Universidad Central del Ecuador; Sandra C Riofrío Terrazas, Dra (c), Study Chair — Centro de Salud San Antonio de Pichincha
Locations (1):
- Centro de Salud de San Antonio de Pichincha, Quito, Pichincha, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang CH, Chung MH, Chan P, Tsai JC, Chen FC. Effects of endurance exercise training on risk components for metabolic syndrome, interleukin-6, and the exercise capacity of postmenopausal women. Geriatr Nurs. 2014 May-Jun;35(3):212-8. doi: 10.1016/j.gerinurse.2014.02.001. Epub 2014 Mar 26. PMID 24679550
- [Result] Lin CH, Chiang SL, Heitkemper MM, Hung YJ, Lee MS, Tzeng WC, Chiang LC. Effects of telephone-based motivational interviewing in lifestyle modification program on reducing metabolic risks in middle-aged and older women with metabolic syndrome: A randomized controlled trial. Int J Nurs Stud. 2016 Aug;60:12-23. doi: 10.1016/j.ijnurstu.2016.03.003. Epub 2016 Mar 12. PMID 27297365
- [Result] Chiang LC, Heitkemper MM, Chiang SL, Tzeng WC, Lee MS, Hung YJ, Lin CH. Motivational Counseling to Reduce Sedentary Behaviors and Depressive Symptoms and Improve Health-Related Quality of Life Among Women With Metabolic Syndrome. J Cardiovasc Nurs. 2019 Jul/Aug;34(4):327-335. doi: 10.1097/JCN.0000000000000573. PMID 30920439
- [Result] Vilchez Barboza V, Klijn TP, Salazar Molina A, Saez Carrillo KL. Effectiveness of personalized face-to-face and telephone nursing counseling interventions for cardiovascular risk factors: a controlled clinical trial. Rev Lat Am Enfermagem. 2016 Aug 8;24:e2747. doi: 10.1590/1518-8345.0626.2747. PMID 27508917
- [Result] Yusuf S, Wood D, Ralston J, Reddy KS. The World Heart Federation's vision for worldwide cardiovascular disease prevention. Lancet. 2015 Jul 25;386(9991):399-402. doi: 10.1016/S0140-6736(15)60265-3. Epub 2015 Apr 16. No abstract available. PMID 25892680
- [Result] Chedraui P, Perez-Lopez FR, Mendoza M, Morales B, Martinez MA, Salinas AM, Hidalgo L. Severe menopausal symptoms in middle-aged women are associated to female and male factors. Arch Gynecol Obstet. 2010 May;281(5):879-85. doi: 10.1007/s00404-009-1204-z. Epub 2009 Aug 14. PMID 19680673
- [Result] Hayman LL, Berra K, Fletcher BJ, Houston Miller N. The Role of Nurses in Promoting Cardiovascular Health Worldwide: The Global Cardiovascular Nursing Leadership Forum. J Am Coll Cardiol. 2015 Aug 18;66(7):864-866. doi: 10.1016/j.jacc.2015.06.1319. No abstract available. PMID 26271070
- [Result] Goncalves JT, Silveira MF, Campos MC, Costa LH. Overweight and obesity and factors associated with menopause. Cien Saude Colet. 2016 Apr;21(4):1145-56. doi: 10.1590/1413-81232015214.16552015. English, Portuguese. PMID 27076013
- [Result] Nunez-Pizarro JL, Gonzalez-Luna A, Mezones-Holguin E, Blumel JE, Baron G, Bencosme A, Benitez Z, Bravo LM, Calle A, Flores D, Espinoza MT, Gomez G, Hernandez-Bueno JA, Martino M, Lima S, Monterrosa A, Mostajo D, Ojeda E, Onatra W, Sanchez H, Tserotas K, Vallejo MS, Witis S, Zuniga MC, Chedraui P. Association between anxiety and severe quality-of-life impairment in postmenopausal women: analysis of a multicenter Latin American cross-sectional study. Menopause. 2017 Jun;24(6):645-652. doi: 10.1097/GME.0000000000000813. PMID 28118294
- [Result] Shin H, Shin HS. Measurement of quality of life in menopausal women: a systematic review. West J Nurs Res. 2012 Jun;34(4):475-503. doi: 10.1177/0193945911402848. Epub 2011 Mar 25. PMID 21441417
- [Result] Sayan S, Pekin T, Yildizhan B. Relationship between vasomotor symptoms and metabolic syndrome in postmenopausal women. J Int Med Res. 2018 Oct;46(10):4157-4166. doi: 10.1177/0300060518790709. Epub 2018 Aug 9. PMID 30092678
- [Result] Zajac-Gawlak I, Klapcinska B, Kroemeke A, Pospiech D, Pelclova J, Pridalova M. Associations of visceral fat area and physical activity levels with the risk of metabolic syndrome in postmenopausal women. Biogerontology. 2017 Jun;18(3):357-366. doi: 10.1007/s10522-017-9693-9. Epub 2017 Mar 18. PMID 28316012
- [Result] Montez JK, Bromberger JT, Harlow SD, Kravitz HM, Matthews KA. Life-Course Socioeconomic Status and Metabolic Syndrome Among Midlife Women. J Gerontol B Psychol Sci Soc Sci. 2016 Nov;71(6):1097-1107. doi: 10.1093/geronb/gbw014. Epub 2016 Feb 28. PMID 26926957
- [Result] Chedraui P, Aguirre W, Hidalgo L, Fayad L. Assessing menopausal symptoms among healthy middle aged women with the Menopause Rating Scale. Maturitas. 2007 Jul 20;57(3):271-8. doi: 10.1016/j.maturitas.2007.01.009. Epub 2007 Feb 27. PMID 17329046
- [Result] Giannouli P, Zervas I, Armeni E, Koundi K, Spyropoulou A, Alexandrou A, Kazani A, Areti A, Creatsa M, Lambrinoudaki I. Determinants of quality of life in Greek middle-age women: a population survey. Maturitas. 2012 Feb;71(2):154-61. doi: 10.1016/j.maturitas.2011.11.013. Epub 2011 Dec 16. PMID 22177978
- [Result] Raczkiewicz D, Owoc A, Wierzbinska-Stepniak A, Bojar I. Metabolic syndrome in peri - and postmenopausal women performing intellectual work. Ann Agric Environ Med. 2018 Dec 20;25(4):610-615. doi: 10.26444/aaem/74451. Epub 2017 Jul 13. PMID 30586981
- [Result] Lee WJ, Yoon JW, Lee JH, Kwag BG, Chang SH, Choi YJ. Effects of Age at First Childbirth and Other Factors on Central Obesity in Postmenopausal Women: The 2013-2015 Korean National Health and Nutrition Examination Survey. Korean J Fam Med. 2018 May;39(3):155-160. doi: 10.4082/kjfm.2018.39.3.155. Epub 2018 May 18. PMID 29788703
- [Result] Kim HR, Kim HS. Optimal Cutoffs of Cardiometabolic Risk for Postmenopausal Korean Women. Asian Nurs Res (Korean Soc Nurs Sci). 2017 Jun;11(2):107-112. doi: 10.1016/j.anr.2017.05.003. Epub 2017 Jun 1. PMID 28688495
- [Result] Tsai SS, Lin YS, Hwang JS, Chu PH. Vital roles of age and metabolic syndrome-associated risk factors in sex-specific arterial stiffness across nearly lifelong ages: Possible implication of menopause and andropause. Atherosclerosis. 2017 Mar;258:26-33. doi: 10.1016/j.atherosclerosis.2017.01.023. Epub 2017 Jan 20. PMID 28182996
- [Result] Mozos I, Malainer C, Horbanczuk J, Gug C, Stoian D, Luca CT, Atanasov AG. Inflammatory Markers for Arterial Stiffness in Cardiovascular Diseases. Front Immunol. 2017 Aug 31;8:1058. doi: 10.3389/fimmu.2017.01058. eCollection 2017. PMID 28912780
- [Result] Miguel-Soca PE, Rivas-Estevez M, Sarmiento-Teruel Y, Marino-Soler AL, Marrero-Hidalgo M, Mosqueda-Batista L, Pena-Perez I, Rivas-Vazquez D, Llorente-Columbie Y. Prevalence of Metabolic Syndrome Risk Factors in Adults in Holguin, Cuba (2004-2013). MEDICC Rev. 2016 Jan-Apr;18(1-2):28. doi: 10.37757/MR2016.V18.N1-2.6. Epub 2016 May 10. No abstract available. PMID 34362239
- [Result] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Result] Aleyasin SA, Navidi T, Davoudi S. Association between rs10757274 and rs2383206 SNPs as Genetic Risk Factors in Iranian Patients with Coronary Artery Disease. J Tehran Heart Cent. 2017 Jul;12(3):114-118. PMID 29062378
- [Result] Hwang YS, Park EJ, Choi JG, Kim HE, Park SG, Yoo SM. Relationship between Age at Menarche and Metabolic Syndrome in Premenopausal Women: Korea National Health and Nutrition Examination Survey 2013-2014. Korean J Fam Med. 2018 Sep;39(5):300-306. doi: 10.4082/kjfm.17.0022. Epub 2018 Jul 30. PMID 30056694
- [Result] Sciomer S, Moscucci F, Dessalvi CC, Deidda M, Mercuro G. Gender differences in cardiology: is it time for new guidelines? J Cardiovasc Med (Hagerstown). 2018 Dec;19(12):685-688. doi: 10.2459/JCM.0000000000000719. PMID 30239478
- [Result] Davis SR, Lambrinoudaki I, Lumsden M, Mishra GD, Pal L, Rees M, Santoro N, Simoncini T. Menopause. Nat Rev Dis Primers. 2015 Apr 23;1:15004. doi: 10.1038/nrdp.2015.4. PMID 27188659
- [Result] Bentley-Lewis R, Koruda K, Seely EW. The metabolic syndrome in women. Nat Clin Pract Endocrinol Metab. 2007 Oct;3(10):696-704. doi: 10.1038/ncpendmet0616. PMID 17893688
- [Result] Oh GC, Kang KS, Park CS, Sung HK, Ha KH, Kim HC, Park S, Ihm SH, Lee HY. Metabolic syndrome, not menopause, is a risk factor for hypertension in peri-menopausal women. Clin Hypertens. 2018 Oct 15;24:14. doi: 10.1186/s40885-018-0099-z. eCollection 2018. PMID 30349737
- [Result] Kozakowski J, Gietka-Czernel M, Leszczynska D, Majos A. Obesity in menopause - our negligence or an unfortunate inevitability? Prz Menopauzalny. 2017 Jun;16(2):61-65. doi: 10.5114/pm.2017.68594. Epub 2017 Jun 30. PMID 28721132
- [Result] Mattei J, Tamez M, Rios-Bedoya CF, Xiao RS, Tucker KL, Rodriguez-Orengo JF. Health conditions and lifestyle risk factors of adults living in Puerto Rico: a cross-sectional study. BMC Public Health. 2018 Apr 12;18(1):491. doi: 10.1186/s12889-018-5359-z. PMID 29650018
- [Result] Sabanovic S, Ljiljana MT, Babic F, Vadovsky M, Paralic J, Vcev A, Holzinger A. Metabolic syndrome in hypertensive women in the age of menopause: a case study on data from general practice electronic health records. BMC Med Inform Decis Mak. 2018 Apr 2;18(1):24. doi: 10.1186/s12911-018-0601-2. PMID 29609615
- [Result] Yeh ML, Liao RW, Hsu CC, Chung YC, Lin JG. Exercises improve body composition, cardiovascular risk factors and bone mineral density for menopausal women: A systematic review and meta-analysis of randomized controlled trials. Appl Nurs Res. 2018 Apr;40:90-98. doi: 10.1016/j.apnr.2017.12.011. Epub 2017 Dec 19. PMID 29579505
- [Result] Oh EG, Bang SY, Kim SH, Hyun SS, Chu SH, Jeon JY, Im JA, Lee JE, Lee MK. Therapeutic lifestyle modification program reduces plasma levels of the chemokines CRP and MCP-1 in subjects with metabolic syndrome. Biol Res Nurs. 2013 Jan;15(1):48-55. doi: 10.1177/1099800411416637. Epub 2011 Aug 22. PMID 21859748
- [Result] Oh EG, Hyun SS, Kim SH, Bang SY, Chu SH, Jeon JY, Kang MS. A randomized controlled trial of therapeutic lifestyle modification in rural women with metabolic syndrome: a pilot study. Metabolism. 2008 Feb;57(2):255-61. doi: 10.1016/j.metabol.2007.09.009. PMID 18191057
- [Result] Beckie TM, Beckstead JW, Groer MW. The influence of cardiac rehabilitation on inflammation and metabolic syndrome in women with coronary heart disease. J Cardiovasc Nurs. 2010 Jan-Feb;25(1):52-60. doi: 10.1097/JCN.0b013e3181b7e500. PMID 19935427
- [Result] Taylor JY, Wu CY. Effects of genetic counseling for hypertension on changes in lifestyle behaviors among African-American women. J Natl Black Nurses Assoc. 2009 Jul;20(1):1-10. PMID 19691178
- [Result] Williams LT, Hollis JL, Collins CE, Morgan PJ. The 40-Something randomized controlled trial to prevent weight gain in mid-age women. BMC Public Health. 2013 Oct 25;13:1007. doi: 10.1186/1471-2458-13-1007. PMID 24156558
- [Result] Williams LT, Hollis JL, Collins CE, Morgan PJ. Can a relatively low-intensity intervention by health professionals prevent weight gain in mid-age women? 12-Month outcomes of the 40-Something randomised controlled trial. Nutr Diabetes. 2014 May 5;4(5):e116. doi: 10.1038/nutd.2014.12. PMID 24799163
- [Result] Lim H, Son JY, Choue R. Effects of medical nutrition therapy on body fat and metabolic syndrome components in premenopausal overweight women. Ann Nutr Metab. 2012;61(1):47-56. doi: 10.1159/000339262. Epub 2012 Jul 20. PMID 22832546
- [Result] Blumenthal JA, Babyak MA, Sherwood A, Craighead L, Lin PH, Johnson J, Watkins LL, Wang JT, Kuhn C, Feinglos M, Hinderliter A. Effects of the dietary approaches to stop hypertension diet alone and in combination with exercise and caloric restriction on insulin sensitivity and lipids. Hypertension. 2010 May;55(5):1199-205. doi: 10.1161/HYPERTENSIONAHA.109.149153. Epub 2010 Mar 8. PMID 20212264
- [Result] Chedraui P, Blumel JE, Baron G, Belzares E, Bencosme A, Calle A, Danckers L, Espinoza MT, Flores D, Gomez G, Hernandez-Bueno JA, Izaguirre H, Leon-Leon P, Lima S, Mezones-Holguin E, Monterrosa A, Mostajo D, Navarro D, Ojeda E, Onatra W, Royer M, Soto E, Tserotas K. Impaired quality of life among middle aged women: a multicentre Latin American study. Maturitas. 2008 Dec 20;61(4):323-9. doi: 10.1016/j.maturitas.2008.09.026. Epub 2008 Nov 17. PMID 19010618